CLINICAL TRIAL: NCT01592409
Title: Acute and Residual Effects of Cannabis on Young Drivers' Performance of Driving-related Skills
Brief Title: Cannabis Effects on Driving-related Skills of Young Drivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Health Canada (Other Government)
Responsible Party: Principal Investigator, Robert Mann, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 125/2011
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Results first posted 2019-02-11 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2018-09

CONDITIONS: Psychomotor Impairment
Keywords: cannabis impaired driving; driving simulation; acute psychopharmacologic effects of cannabis; residual effects of cannabis; young drivers
MeSH Terms: conditions — Psychomotor Disorders | interventions — Dronabinol; nabiximols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active cannabis (Active Comparator): In this condition, participants will receive a cigarette containing 12.5% active THC.
  Interventions: Drug: delta-9-tetrahydrocannabinol
- Placebo (Placebo Comparator): In this condition, participants will receive a cannabis cigarette where the active THC has been removed (contains 0% THC).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: delta-9-tetrahydrocannabinol — A single cannabis cigarette (potency 12.5% THC) will be given to participants to smoke over a 10 minute period, ad lib. If the cigarette is not smoked in its entirety, the remainder will be weighed to estimate dose.
  Other Names: cannabis sativa; marijuana
  Arms: Active cannabis
Drug: Placebo — A single placebo cannabis cigarette (0% THC) will be given to participants to smoke over a 10 minute period, ad lib. If the cigarette is not smoked in its entirety, the remainder will be weighed to estimate dose (as this is a double-blind study).
  Other Names: cannabis sativa; marijuana
  Arms: Placebo

SUMMARY:
Motor vehicle collisions are the leading cause of death for young people. The investigators have recently found that driving after using cannabis is more common among young Canadian drivers than driving after drinking. While this observation raises concerns, the effects of cannabis on driving-related skills in this age group are not well understood. As well, evidence suggests that residual effects of cannabis on driving-related skills may be observed up to 24 hours later. These residual effects may have important implications for the effects of cannabis use on collision risk, but little evidence on them in available. This study will examine the effects of a single dose of cannabis (marijuana) on driving-related skills immediately following consumption, 24 hours later, and 48 hours later. To date, the residual effect at 48 hours has not been examined. A total of 142 subjects aged 19 to 25 years old will be randomly assigned to smoke either a placebo or active cannabis cigarette (12.5% THC potency). Following an eligibility screening and practice session, participants will attend 3 testing days; drug-administration, 24-hour follow-up and 48-hour follow-up. The effects of cannabis/placebo on performance of driving-related skills using a high-fidelity driving simulator will be assessed on each testing day. The effects of cannabis on mood, cognition, memory and complex reaction time will also be assessed. Identifying factors that affect the collision risks experienced by young drivers is a public health priority. While many young people believe that cannabis does not impair driving, some recent studies suggest that these may be very dangerous beliefs. This study will provide important information on how cannabis may affect the driving skills of young drivers, to inform efforts to understand and address cannabis-related collision in this age group.

DETAILED DESCRIPTION:
This study will test the prediction that residual effects of an acute dose of cannabis on driving-related skills will be observed in a group of young drivers 48 hours following a single dose of smoked cannabis, and will also examine the effects of an acute dose of cannabis on those skills using driving simulator technology.

Study Objectives

1. Examine the residual effects of a moderate dose of cannabis (12.5% THC) on driving simulator performance of young drivers. Simulated driving performance, tests of cognition, verbal memory, and mood will be measured concurrently with levels of cannabinoids in biological fluids at approximately 24 and 48 hours following acute drug exposure in male and female drivers aged 19 to 25. We will test the hypothesis that performance on a high-fidelity driving simulator task will be significantly impaired approximately 24 hours following a dose of cannabis in comparison to a placebo condition.
2. Examine the acute effects of a moderate dose of cannabis (12.5% THC) on driving simulator performance of young drivers. Simulated driving performance, tests of cognition, verbal memory, and mood will be measured concurrently with levels of cannabinoids in biological fluids before and after drug administration. Cannabinoid levels in biological fluids will be measured over a 6 hour period following drug exposure. We will examine the relationship of cannabinoid levels to performance measures in this time frame.
3. Explore the effects of driving history, driving attitudes, and individual difference measures (e.g., demographics, drug and alcohol use, etc.) on the acute and residual effects of cannabis on driving simulator performance of young drivers. Exploratory analyses will be undertaken to determine if the acute and residual effects of cannabis on the driving simulator task are influenced by these measures.
4. Determine if a relationship exists between genetics and THC response. As an ancillary aim, blood samples may be collected for future research to determine if a relationship exists between genetic polymorphisms and pharmacokinetic and pharmacodynamic responses to cannabis.

Study Design and Duration

The study is a double-blind, placebo-controlled mixed-design study, including a randomized between-subjects comparison of the effects of smoked cannabis and both between- and within-subjects examination of its residual effects at 24 and 48 hours following one-time drug administration. Although a placebo condition is part of the study, this is not a treatment study.

Initial contact with potential subjects will be made via telephone, and study personnel will conduct a telephone screen for eligibility. Upon eligibility confirmation by telephone, participants will be asked to attend CAMH for an eligibility assessment. The study will consist of 5 sessions for each subject (an eligibility assessment, a practice day, and three subsequent testing days). Participants will be asked not to use cannabis for 48 hours prior to attending the practice day (Session 2). Although Session 1 can be completed at any time prior to the remaining study sessions, Sessions 2 - 5 must be performed on consecutive days.

In certain instances, the Qualified Investigator may ask a participant to return for re-screening, e.g. repeat of urine test or other assessments performed for eligibility assessment. Also, in case of unforeseen delays in scheduling study participation, the Qualified Investigator will determine if there is a need to ask a participant to repeat some assessments, e.g., physical examination.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 19 to 25
* Regular cannabis users (between one and four times per week)
* Held a valid class G or G2 Ontario driver's license (or equivalent from another jurisdiction) for at least 12 months.
* Willing to abstain from cannabis use for the duration of the study, and for 48 hours prior to Session 2.
* Provides written and informed consent
* Urine toxicology result positive for THC (indicating recent use of cannabis).

Exclusion Criteria:

* Positive breathalyzer results for alcohol on any given study day.
* Is a regular user of medications that affect brain function (i.e., antidepressants, benzodiazepines, stimulants).
* Diagnosis of severe medical or psychiatric conditions.
* A first degree relative diagnosed with schizophrenia.
* Meets criteria for current or lifetime Substance Use Disorders (DSM-IV) with the exception of nicotine.
* Meets criteria for Cannabis Dependence (DSM-IV).
* Is pregnant, is trying to become pregnant, or is currently breastfeeding.

Ongoing Exclusion Criteria:

* Upon eligibility assessment, toxicology results indicate that the participant has not used cannabis recently.
* Any toxicology screen after Session 2 - Practice Day indicating a psychoactive substance has been used other than cannabis.

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2012-07; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Mann, Ph.D., Principal Investigator — Centre for Addiction and Mental Health; Bernard Le Foll, M.D., Ph.D., Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Background] Adlaf EM, Begin P, Sawka E. Canadian Addiction Survey (CAS): A national survey of Canadians' use of alcohol and other drugs: Prevalence of use and related harms: Detailed report. Ottawa, Canada: Canadian Cenre for Substance Abuse 2005
- [Background] Johnston LD, O'Malley PM, Backman JG, Schulenber JE. Monitoring the future: National results on adolescent drug use. Bethesda, MD.: National Institute on Drug Abuse 2009
- [Background] WHO - Programme on substance abuse. Cannabis: a health perspective and research agenda: World Health Organization 1997.
- [Background] Chipman ML, Macdonald S, Mann RE. Being "at fault" in traffic crashes: does alcohol, cannabis, cocaine, or polydrug abuse make a difference? Inj Prev. 2003 Dec;9(4):343-8. doi: 10.1136/ip.9.4.343. PMID 14693897
- [Background] Brault M, Dussault C, Bouchard J, Lemire AM. The contribution of alcohol and other drugs among fatally injured drivers in Quebec: final results. Société de l'assurance automobile du Quebec 2002. Available from: http://www.saaq.gouv.qc.ca/publications/dossiers_etudes/drogue_an.pdf
- [Background] Laumon B, Gadegbeku B, Martin JL, Biecheler MB; SAM Group. Cannabis intoxication and fatal road crashes in France: population based case-control study. BMJ. 2005 Dec 10;331(7529):1371. doi: 10.1136/bmj.38648.617986.1F. Epub 2005 Dec 1. PMID 16321993
- [Background] Siliquini R, Chiado Piat S, Gianino MM, Renga G. Drivers involved in road traffic accidents in Piedmont Region: psychoactive substances consumption. J Prev Med Hyg. 2007 Dec;48(4):123-8. PMID 18557306
- [Background] Stoduto G, Vingilis E, Kapur BM, Sheu WJ, McLellan BA, Liban CB. Alcohol and drug use among motor vehicle collision victims admitted to a regional trauma unit: demographic, injury, and crash characteristics. Accid Anal Prev. 1993 Aug;25(4):411-20. doi: 10.1016/0001-4575(93)90070-d. PMID 8357454
- [Background] Drummer OH, Gerostamoulos J, Batziris H, Chu M, Caplehorn J, Robertson MD, Swann P. The involvement of drugs in drivers of motor vehicles killed in Australian road traffic crashes. Accid Anal Prev. 2004 Mar;36(2):239-48. doi: 10.1016/s0001-4575(02)00153-7. PMID 14642878
- [Background] Lacey JH, Kelley-Baker T, Furr-Holden D, Voas RB, Romano E, Ramirez A, et al. 2007 National roadside survey of alcohol and drug use by drivers: Drug results. Washington, DC: National Highway Traffic Safety Administration 2009.
- [Background] Blows S, Ivers RQ, Connor J, Ameratunga S, Woodward M, Norton R. Marijuana use and car crash injury. Addiction. 2005 May;100(5):605-11. doi: 10.1111/j.1360-0443.2005.01100.x. PMID 15847617
- [Background] Asbridge M, Poulin C, Donato A. Motor vehicle collision risk and driving under the influence of cannabis: evidence from adolescents in Atlantic Canada. Accid Anal Prev. 2005 Nov;37(6):1025-34. doi: 10.1016/j.aap.2005.05.006. Epub 2005 Jun 29. PMID 15992751
- [Background] Adlaf EM, Mann RE, Paglia A. Drinking, cannabis use and driving among Ontario students. CMAJ. 2003 Mar 4;168(5):565-6. PMID 12615749
- [Background] Fischer B, Rodopoulos J, Rehm J, Ivsins A. Toking and driving: Characteristics of Canadian university students who drive after cannabis use - an exploratory pilot study. Drugs Ed Prev Policy 13:179-87, 2006
- [Background] O'Malley PM, Johnston LD. Drugs and driving by American high school seniors, 2001-2006. J Stud Alcohol Drugs. 2007 Nov;68(6):834-42. doi: 10.15288/jsad.2007.68.834. PMID 17960301
- [Background] McGuire F, Dawe M, Shield KD, Rehm J, Fishcher B. Driving under the influence of cannabis or alcohol in a cohort of high-frequency cannabis users: prevalence and reflections on current interventions. Canadian Journal of Criminology and Criminal Justice 53(2): 247-259, 2011
- [Background] Pope HG Jr, Gruber AJ, Yurgelun-Todd D. The residual neuropsychological effects of cannabis: the current status of research. Drug Alcohol Depend. 1995 Apr;38(1):25-34. doi: 10.1016/0376-8716(95)01097-i. PMID 7648994
- [Background] Heishman SJ, Huestis MA, Henningfield JE, Cone EJ. Acute and residual effects of marijuana: profiles of plasma THC levels, physiological, subjective, and performance measures. Pharmacol Biochem Behav. 1990 Nov;37(3):561-5. doi: 10.1016/0091-3057(90)90028-g. PMID 1965045
- [Background] Smiley A. Marijuana: On-road and driving simulator studies. Alcohol, Drugs, and Driving. 2:121-34, 1986
- [Background] Crancer A Jr, Dille JM, Delay JC, Wallace JE, Haykin MD. Comparison of the effects of marihuana and alcohol on simulated driving performance. Science. 1969 May 16;164(3881):851-4. doi: 10.1126/science.164.3881.851. PMID 5767792
- [Background] Cone EJ, Huestis MA. Relating blood concentrations of tetrahydrocannabinol and metabolites to pharmacologic effects and time of marijuana usage. Ther Drug Monit. 1993 Dec;15(6):527-32. doi: 10.1097/00007691-199312000-00013. PMID 8122288
- [Background] Harder S, Rietbrock S. Concentration-effect relationship of delta-9-tetrahydrocannabiol and prediction of psychotropic effects after smoking marijuana. Int J Clin Pharmacol Ther. 1997 Apr;35(4):155-9. PMID 9112136
- [Background] McLaren J, Swift W, Dillon P, Allsop S. Cannabis potency and contamination: a review of the literature. Addiction. 2008 Jul;103(7):1100-9. doi: 10.1111/j.1360-0443.2008.02230.x. Epub 2008 May 20. PMID 18494838
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collaborating Centre — http://www.camh.net/research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was by media ads and research postings in Toronto.
Pre-assignment Details: Screened over the telephone n=1024. Assessed for eligibility (n=178). Excluded: Not meeting inclusion criteria n=45, Declined to participate or lost interest n=32, Did not receive IP (did not return after practice session) n=2.
  Pilots (received active cannabis, not randomized) n=5. Randomized n=94.
Period: Overall Study
Arm/Group | Active Cannabis | Placebo
Started | 67 | 32
Completed | 67 | 31
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: One participant was excluded from analyses because they admitted to having tried to skew their data. They withdrew from the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Cannabis | Placebo | Total
Number analyzed (Participants) | 67 | 31 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.22 (1.88) | 21.97 (2.24) | 22.14 (1.995)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 9 | 28
  Male | 48 | 22 | 70
Region of Enrollment [Number; unit: participants]
  Canada | 67 | 31 | 98

OUTCOME MEASURES:

1. Primary Outcome: Psychomotor Impairment (Driving)
Description: The driving simulator will objectively measure driving behaviour during a number of pre-programmed driving scenarios. Zone/ Hazard performance measure: Mean Speed.
Time Frame: Approximate: at baseline (30 minutes before smoking), 30 minutes after smoking
Population: Zone/Hazard performance measure: Mean Speed (Change from drug-free baseline to 30 minutes after smoking cannabis in kilometres per hour (kph)
Measure: Mean (Standard Deviation); unit: change in kph
Arm/Group | Active Cannabis | Placebo
Number analyzed (Participants) | 67 | 31
change in kph | 3.38 (9.75) | -1.54 (7.36)

ADVERSE EVENTS:
Time Frame: Collected from session 1 (eligibility assessment) to session 2 (practice) (approx. 3 months); from session 2 to 3 (approx. 24 hours), from session 3 to 4 (approx. 24 hours), session 4 to session 5 (approx. 24 hours).
Arm/Group | Active Cannabis | Placebo
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/32
Other Adverse Events (participants affected / at risk) | 38/67 | 15/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Cannabis (N=67) | Placebo (N=32)
injury (Musculoskeletal and connective tissue disorders) | 0 | 2 — sprained ankle, burn
bruising (Skin and subcutaneous tissue disorders) | 1 | 1 — at site of blood draw
allergies (Immune system disorders) | 0 | 1
anxiety/nervousness (Psychiatric disorders) | 1 | 2
common cold (Respiratory, thoracic and mediastinal disorders) | 3 | 1
dizziness/faintness (General disorders) | 5 | 2
diaphoresis (General disorders) | 1 | 0
difficulty falling asleep (General disorders) | 1 | 0
genital discomfort (Reproductive system and breast disorders) | 1 | 1
headache (General disorders) | 10 | 2
earache (Ear and labyrinth disorders) | 1 | 0
food poisoning (Gastrointestinal disorders) | 1 | 0
insomnia (General disorders) | 6 | 0
increased appetite (Metabolism and nutrition disorders) | 0 | 1
low blood pressure (Vascular disorders) | 4 | 1
itching (Skin and subcutaneous tissue disorders) | 1 | 0
loss of consciousness (Vascular disorders) | 2 | 0 — vasovagal episode
muscle/bone/joint pain (Musculoskeletal and connective tissue disorders) | 3 | 2 — arm
nausea (Gastrointestinal disorders) | 1 | 1
nasal infection (General disorders) | 1 | 0
rapid heartbeat (Cardiac disorders) | 2 | 0
rash (Skin and subcutaneous tissue disorders) | 4 | 0
simulation sickness (Ear and labyrinth disorders) | 1 | 2 — nausea/dizziness due to driving simulator
somnolence (General disorders) | 4 | 1
sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
stomach/abdominal discomfort (Gastrointestinal disorders) | 2 | 0
tiredness/fatigue (General disorders) | 5 | 3
vomiting (Gastrointestinal disorders) | 0 | 1
abdominal pain (Gastrointestinal disorders) | 3 | 0

LIMITATIONS AND CAVEATS:
The study examined simulated driving behavior of young regular cannabis users (1 to 4 times per week) and the generalization to new or frequent cannabis users, older drivers, and to real-world driving is unclear.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes